CLINICAL TRIAL: NCT06754423
Title: Electronic Registry of Male Patients With Congenital Adrenal Hyperplasia 21-hydroxylase Deficiency
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: AndroCAH
Record Dates: First submitted 2024-12-01; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Congenital Adrenal Hyperplasia
Keywords: Congenital adrenal hyperplasia
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Observational, retrospective, prospective, single-center cohort study. Participation in the registry will be offered consecutively to any patient with the disease, newly diagnosed or with documented diagnosis made at another center, at any stage of the disease. Laboratory tests, imaging study for patient monitoring and care procedures all will be conducted in accordance with normal clinical practice.

DETAILED DESCRIPTION:
Observational, retrospective, prospective, single-center cohort study conducted at the UOC of Endocrinology and Diabetes Prevention and Treatment of IRCCS AOU of Bologna. Participation in the Registry will be offered consecutively to any patient with the disease, newly diagnosed or with documented diagnosis made at another Center, at any stage of the disease. Laboratory tests, imaging study for patient monitoring, and care procedures all will be conducted in accordance with normal clinical practice.

For the retrospective phase, patients whose diagnosis of CAH was made on or after 01/01/1960 will be enrolled, and observation related to this phase will be extended until this study is approved.

The study population is partly from direct access at the U.O.C. of Endocrinology and Diabetes Prevention and Treatment, as the regional referral center for this rare disease (congenital adrenal hyperplasia).

The potentially involved cohort is estimated to be about 30 patients at the time the registry was established. It is assumed that both retrospective and prospective phases can be completed in 15 subjects and retrospective alone in the remaining 15 subjects.

The registry may become the reference for calculating incidence and prevalence in Emilia Romagna of the disease under study.

ELIGIBILITY:
Inclusion Criteria:

* Male gender;
* Age 18 years or older;
* Newly or previously diagnosed patients with CAH from 21-hydroxylase enzyme deficiency, in whom CYP21A2 gene analysis for determination of pathological mutations and genotype has already been performed;
* Obtaining informed consent.

Exclusion Criteria:

* Patients with an unsure diagnosis of CAH;
* Patients with CAH caused by (or with the co-presence of) pathogenic molecular alterations other than mutations in the CYP21A2 gene.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male gender
Study Population: The study population partly comes from direct access at the O.U. of Endocrinology and Diabetes Prevention and Treatment, as a regional referral center for this rare disease (congenital adrenal hyperplasia). A second part afferents instead from the O.U. of Pediatrics of the Polyclinic through the "interdepartmental procedure for the management of the transition of patients with endocrine-metabolic diseases from pediatric endocrinology to adult endocrinology."
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-06-24 (Actual); Primary Completion 2032-06-24 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Creation of an electronic registry | through study completion, an average on 31 December 2032
  The primary objective of the study is to create an electronic registry and, through the data contained therein, to describe the clinical-laboratory aspects, prevalence, and type of alterations in gonadal function of a cohort of male patients, aged 18 years or older, with congenital adrenal hyperplasia from 21-hydroxylase deficiency regardless of the time of diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Gambineri, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero Universitaria di Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No